CLINICAL TRIAL: NCT01212887
Title: A Cancer Research UK Phase I Trial of Adoptive Transfer of Autologous Tumor Antigen-Specific T Cells With Preconditioning Chemotherapy and Intravenous IL2 in Patients With Advanced CEA Positive Tumors
Brief Title: Treated Blood Cells, Cyclophosphamide, Fludarabine Phosphate, and Aldesleukin in Treating Patients With Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to safety concerns and lack of efficacy
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000685060; CRUK-PH1/105; CRUK-MFEz; EUDRACT-2005-004085-16; EU-21070
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Gastric Cancer; Lung Cancer; Ovarian Cancer; Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent colon cancer; stage IIIA colon cancer; stage IIIB colon cancer; stage IIIC colon cancer; stage IV colon cancer; stage IVB colon cancer; recurrent rectal cancer; stage IIIA rectal cancer; stage IIIB rectal cancer; stage IIIC rectal cancer; stage IVA rectal cancer; stage IVB rectal cancer; recurrent gastric cancer; stage IV gastric cancer; recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent breast cancer; stage IIIC breast cancer; stage IV breast cancer; extensive stage small cell lung cancer; recurrent non-small cell lung cancer; recurrent small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage IIIA ovarian epithelial cancer; stage IIIA ovarian germ cell tumor; stage IIIB ovarian epithelial cancer; stage IIIB ovarian germ cell tumor; stage IIIC ovarian epithelial cancer; stage IIIC ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Ovarian Epithelial | interventions — aldesleukin; Cyclophosphamide; fludarabine phosphate

INTERVENTIONS:
Biological: MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes
Biological: aldesleukin
Drug: cyclophosphamide
Drug: fludarabine phosphate
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Placing a gene into T cells may improve the body's ability to recognize cancer cells and build an immune response to fight cancer. Drugs used in chemotherapy, such as cyclophosphamide and fludarabine phosphate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Biological therapies, such as aldesleukin, may stimulate the immune system in different ways and stop cancer cells from growing. Giving specially treated T cells together with cyclophosphamide, fludarabine phosphate, and aldesleukin may kill more tumor cells.

PURPOSE: This phase I clinical trial is studying the side effects and best dose of treated T cells when given together with cyclophosphamide, fludarabine phosphate, and aldesleukin in treating patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the feasibility of MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes in combination with preconditioning chemotherapy comprising cyclophosphamide and fludarabine phosphate plus aldesleukin in patients with CEA-positive tumors.
* To assess the toxicity of this regimen in these patients.
* To determine the dose of MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes required to give optimal survival of these cells in the circulation (recommended phase II dose).

Secondary

* To assess whether MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes isolated from the circulation are functional.
* To determine the preliminary tumor response to MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes.
* To evaluate the safety of MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes.

OUTLINE: This is a phase I, dose-escalation study of MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes.

Patients undergo leukapheresis 7-14 days before study therapy begins. Cells are then transduced with a retrovirus vector and expanded to produce MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes.

Patients receive preconditioning chemotherapy comprising fludarabine phosphate IV over 15 minutes on days -5 to -1 or cyclophosphamide IV over 1 hour on days -7 to -6 and fludarabine phosphate IV over 15 minutes on days -5 to -1. They receive MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes IV over 30 minutes on day 0. Patients also receive high-dose aldesleukin IV over 15 minutes every 8 hours for up to 12 doses beginning on day 0, in the absence of disease progression or unacceptable toxicity. If there is evidence of MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes survival, patients may receive additional high-dose aldesleukin.

Patients undergo blood sample collection periodically for pharmacokinetic and pharmacodynamic studies. Some patients may undergo a tumor biopsy.

After completion of study treatment, patients are followed up every 2 weeks for 6 weeks, every 4 weeks for 6 months, every 3 months for 1 year, and then every 6 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy

  * Metastatic or unresectable disease
  * Standard curative or palliative measures do not exist, are no longer effective, have been completed, or have been refused
* CEA-positive tumor (either by immunohistochemistry or as demonstrated by elevated CEA > 50 μg/L)
* No primary brain tumor or brain metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy ≥ 3 months
* Hemoglobin ≥ 10 g/dL
* Platelet count ≥ 100 x 10^9/L
* Neutrophil count ≥ 2.0 x 10^9/L
* Lymphocyte count ≥ 1.0 x 10^9/L
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT/AST ≤ 5 times ULN
* Alkaline phosphatase ≤ 5 times ULN
* Calculated creatinine clearance OR isotope clearance measurement ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 4 weeks prior to, during, and for 6 months after completion of study therapy (male patients must use barrier-method contraception)
* LVEF ≥ 50% on MUGA scan (for patients receiving cyclophosphamide)
* ECG and exercise ECG (or stress ECHO) normal (may be abnormal but not clinically significant)
* Urine dipstick normal (may be abnormal but not clinically significant)
* No medical high risk due to nonmalignant systemic disease including active uncontrolled infection
* No known serologically positive hepatitis B, hepatitis C, HIV, or HTLV
* No history of autoimmune disease
* No inflammatory bowel disease
* No concurrent congestive heart failure or prior history of NYHA class III-IV cardiac disease
* No concurrent malignancies originating from other primary sites, except for adequately treated cone-biopsied carcinoma in situ of the cervix uteri or basal cell or squamous cell carcinoma of the skin
* No other condition that, in the investigator's opinion, would make the patient an unsuitable candidate for the clinical trial

PRIOR CONCURRENT THERAPY:

* At least 30 days since prior and no concurrent participation in another clinical trial
* At least 4 weeks since prior and no concurrent radiotherapy (except for palliative reasons [i.e., control of bone pain])
* At least 4 weeks since prior and no concurrent endocrine therapy, immunotherapy, or chemotherapy (6 weeks for nitrosoureas and mitomycin C)
* No toxic manifestations of previous treatment, except for alopecia or certain grade 1 toxicities that, in the opinion of the investigator and CRUK (Cancer Research UK), would exclude the patient (e.g., grade 1 neuropathy or grade 1 fatigue)
* No prior major thoracic and/or abdominal surgery from which the patient has not yet recovered
* No prior bone marrow transplant or extensive radiotherapy to > 25% of bone marrow
* No concurrent systemic steroids or other immunosuppressive therapy
* No other concurrent anticancer therapy or investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients (goal is 50%) who are evaluable for MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes survival
Adverse event according to CTCAE version 3 criteria
Dose of MFE23 scFv-expressing autologous anti-CEA MFEz T lymphocytes that gives the highest frequency in the circulation as measured by the primary assays (recommended phase II dose)

SECONDARY OUTCOMES:
Presence of cells with a functional chimeric immune receptor on bCEA binding assay
Partial response or complete response on CT scans at 6, 12, 24, and 52 weeks as defined by RECIST criteria
Long-term follow up for insertional mutagenesis

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Hawkins, MD, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital, Manchester, England, United Kingdom